CLINICAL TRIAL: NCT07102992
Title: Post Burn Cubital Tunnel Syndrome Response to High Intensity Laser Therapy Versus Shock Wave Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud H Mohamed, PhD, Associate Professor, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HILT-SHWT 2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Post Burn Cubital Tunnel Syndrome
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized controlled trial with 3 arms receiving different interventions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity laser therapy (Experimental): Device: High intensity laser therapy 25 Patients
  Interventions: Device: High intensity laser therapy; Other: Ulnar nerve gliding exercises.
- Shock Wave therapy (Active Comparator): Extracorporeal shock wave therapy, 25 patients
  Interventions: Device: Shock Wave therapy; Other: Ulnar nerve gliding exercises.
- Ulnar nerve gliding exercises. (Active Comparator): Ulnar nerve gliding exercises, 25 patients
  Interventions: Other: Ulnar nerve gliding exercises.

INTERVENTIONS:
Device: High intensity laser therapy — High intensity Laser Therapy :A standard handpiece endowed with fixed spacers will used to provide the same distance to the skin and perpendicularly to the zone to be treated with a laser beam diameter of 5 mm. Three phases of treatment will be performed for every session. The total energy that will be delivered to the patient during one session will be 1275 J through three phases of treatment.
  Frequency of treatment: Treatment will be given 5 times / week for 20 sessions.
  Arms: High intensity laser therapy
Device: Shock Wave therapy — radial extracorporeal shock wave therapy (2,000 shots, 4 Bar, 5 Hz) (once a week) will be administered to the ulnar nerve at the proximal cubital tunnel region.
  Frequency of treatment: Treatment will be given 1 time / week for 4 sessions
  Arms: Shock Wave therapy
Other: Ulnar nerve gliding exercises. — While keeping patients head in a neutral position, will teach the patient to:
  1. Begin with your arm out, palm side of the hand facing up.
  2. Bend the elbow toward you, palm side facing you.
  3. Rotate the palm of your hand outward and bend your wrist so that the fingers are pointing towards you.
  4. Twist your wrist so that the palm of your hand is now facing upward.
  5. While your wrist remains bent, stretch out your arm into a straight position, with your fingers bent towards the floor.
  Hold each position for 5 seconds, repeat series 3-5 times. Frequency of treatment: Treatment will be given 5 times / week for 20 sessions.
  Other Names: Ulnar nerve gliding exercises

SUMMARY:
Significant morbidity in burn patients occurs frequently because of Post burn nerve entrapment syndromes. Nerve entrapment arises due to direct compression because of edema; they may also present due to scar tissue formation.

Burns of the forearm and elbow are associated with swelling, redness and pain. In second to third-degree burns, the eschar forms a tight band constricting the circulation distally and forms edema that leads to compression neuropathy of ulnar nerve. Also the hyper metabolic response of the burned patients, has been suggested as a cause of the peripheral neuropathies, as the basal metabolic rate (B.M.R) of the burned patients increase more than 2 to 2.5 times normal.

DETAILED DESCRIPTION:
Significant morbidity in burn patients occurs frequently because of Post burn nerve entrapment syndromes. Nerve entrapment arises due to direct compression because of edema; they may also present due to scar tissue formation.

Burns of the forearm and elbow are associated with swelling, redness and pain. In second to third-degree burns, the eschar forms a tight band constricting the circulation distally and forms edema that leads to compression neuropathy of ulnar nerve. Also the hyper metabolic response of the burned patients, has been suggested as a cause of the peripheral neuropathies, as the basal metabolic rate (B.M.R) of the burned patients increase more than 2 to 2.5 times normal.

Cubital tunnel syndrome is the second most common entrapment neuropathy of the upper extremity, after carpal tunnel syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years.
2. Both sexes.
3. Post healed elbow burn.
4. Diagnosed with cubital tunnel syndrome.
5. Willing and able to provide informed consent.

Exclusion Criteria:

1. Patients with brachial plexopathy.
2. C8-T1 radiculopathy, polyneuropathy.
3. Previous elbow fractures or operation.
4. Systemic diseases such as diabetes mellitus, malignancy, and active infection.
5. Patients with any contraindications to high intensity laser therapy or shock wave therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Nerve Conduction Studies of ulnar nerve | Baseline and 4 weeks
  Nerve conduction studies will assess the function/integrity of the ulnar nerve. Patients will be evaluated at base line before treatment and after completion of treatment using Neuropack S1MEB-9004 NIHON KODEN, JAPAN for measuring the motor conduction velocity of the ulnar nerve.

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Baseline and 4 weeks
  The DASH questionnaire consists of 30 questions regarding limitations to complete physical activities due to upper extremity pain/impairment. Participants will be asked to respond to each question based on their experiences over the preceding week according to a 5-point Likert scale ranging from
  1 (no difficulty) to 5 (unable to do). Responses will be scored out of 5 and averaged to produce a score out of 100 with higher scores representing greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Mansour, Ph.D, Study Chair — Faculty of Physical Therapy, Benha university
Locations (2):
- Egypt (2):
  - Out patient clinic , faculty of Physical Therapy, Benha university, Banhā, Al Qalyubia
  - Out patient clinic , faculty of Physical Therapy, ahram Canadian university, Giza, Giza Governorate

IPD SHARING:
Plan to Share IPD: Undecided